CLINICAL TRIAL: NCT02001961
Title: Using Novel Blood and Imaging Biomarkers to Better Understand the Pathophysiology of Paediatric Dilated Cardiomyopathy
Brief Title: Pathophysiology of Dilated Cardiomyopathy
Status: Withdrawn | Type: Observational
Why Stopped: Study was withdrawn prior to R&D approval
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 12CC23
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Dilated Cardiomyopathy
Keywords: Fibrosis; collagen metabolism; paediatric, dilated cardiomyopathy; biomarkers; T1 mapping; MRI
MeSH Terms: conditions — Cardiomyopathy, Dilated; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma (>400 UL) will be collected in heparinised tubes plasma will be extracted and the cell fraction discarded. Plasma will be stored at 80°C prior to transport on dry ice, via protected courier.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heart failure: Patients will be recruited from the heart failure clinic by their consultant. These will include patients who are due to have a MRI scan for clinical reasons and those who volunteer to participate. Voluntary subjects will be over 8 years.
- Control: Control subjects will be identified after being referred for an MRI scan and being allocated to a non-cardiac MRI with gadolinium contrast.

SUMMARY:
This will be a cross-sectional, observational study.

Null hypothesis:

There is no difference in the amount of extracellular volume (ECV or scarring) in the hearts of patients with heart failure as compared to control subjects.

Heart failure occurs when the heart muscle has become too weak to work properly. It is associated with an increase in the amount of connective tissue (collagen) which replaces dead heart muscle cells (scarring). Currently a biopsy of the muscle is the only way to measure the amount of scarring. This is invasive and rarely done in children. Because of this, it is difficult to measure the amount of scarring in a particular patient or disease process, which is important for improving our understanding and treatment of the disease.

Cardiac magnetic resonance imaging (MRI) is a non-invasive imaging tool which is routinely used to look at areas of local scarring in heart muscle. Because the scarring is so widespread in paediatric patients, we have not been able to use this method previously. Now new imaging techniques allow us to look at widespread scarring but these have not yet been validated in children.

We plan to use late gadolinium enhancement (T1 mapping) to measure the amount of scarring in patients with heart failure (we have evidence that their heart biopsies show increased amounts of scar tissue) and children having MRI scans for other reasons. We will use measures of function including echocardiography and 6 minute walk test to compare to the amount of scarring. This will help us to know whether the amount of scarring will be clinically useful.

We will look at the amount of various proteins in the blood of patients and control subjects which are related to the scarring and cell death processes. We already use blood tests to monitor heart failure and these tests may help us to refine our testing and improve timing of treatment (e.g. transplantation).

This study will help us to design further research in this field.

DETAILED DESCRIPTION:
All patients will be under the care of Great Ormond Street Hospital.

Patient Groups:

There will be three main patient groups:

1. Heart Failure Patients (MRI Clinically indicated)
2. Heart Failure Patients (Voluntarily recruited from clinic)

   1. 8-16 years of age
   2. Non-GA only
3. Control subjects (Clinically indicated brain MRI with contrast)

Patient recruitment

We will include Great Ormond Street patients in this trial who are known to the heart failure team because they have been diagnosed with DCM for at least 3 months. They will have an established diagnosis of heart failure and will be under regular follow up. Where possible, we will attempt to align the research study review date with that of the patient's regular annual review.

We will include patients who are to have a cardiac MRI scan with contrast for clinical reasons. These patients will be of any age and will have the scan under GA if appropriate, In addition, we will recruit patients from heart failure clinic who are not due to have scans for clinical reasons. These patients will be between 8-16 years to allow cooperation with the MRI scan protocol without the need for general anaesthetic (GA).

Age-matched control patients will be those having routine MRI with contrast for non-cardiac MRI scans. They will also have blood tests for cardiac biomarkers at the time of insertion of the cannula for contrast injection. These will be patients identified as requiring gadolinium contrast for neurological imaging. They will include patients who are awake and those sedated or under GA. These patients will mainly be having routine brain MRI with contrast for epilepsy.

Both groups will be fully consented.

Heart Failure Patients:

We will recruit patients being referred for cardiac MRI scanning for clinical reasons as well as inviting patients to volunteer for an MRI. Patients who do not require a cardiac MRI for clinical reasons will be over the age of 8 years to allow for cooperation with the MRI without general anaesthesia. Patients under follow up by the heart failure team will be contacted by their primary care consultant in the first instance to introduce the study and invite the patient to participate. It will be made clear there is no obligation to join the study and their treatment will be unaffected by their decision. They will be free to withdraw consent at any time. The patients will be invited to phone the study coordinator (DP) to ask questions, express willingness to participate or to decline. Non-responders will be sent one further letter of invitation.

Control subjects:

Patients being referred to the MRI department at Great Ormond Street Hospital will be identified once they have been allocated to a neurological MRI protocol with gadolinium enhancement. The radiologist allocating the patient will contact the patients' primary consultant to inform them about the study and request permission to contact the family. The family will be contacted once permission has been given, first by phone and then information sheets will be provided. The patients will be invited to phone the study coordinator (DP) to ask questions, express willingness to participate or to decline. Non-responders will be sent one further letter of invitation.

Travel costs will be reimbursed where these are incurred specifically for participation in the study.

Consent:

Written, informed consent will be obtained from all participants if they choose to take part in this study. Information sheets will also be provided to the patients' GP and their cardiology physician, if they are under separate cardiology follow-up. Patients will be free to withdraw at any time.

Risks & Burdens from the study protocol

The main risk arising from our study relates to the insertion of an IV line and administration of a gadolinium-based contrast agent. Such contrast agents are widely used in clinical practice and are extremely safe when administered within standard dosage guidelines. There are, however, potential complications of allergic reaction and development of Nephrogenic Systemic Fibrosis (NSF). Such allergic reactions are rare and when they occur, the majority are mild.

To mitigate this risk we will exclude patients with a previous history of allergic response to gadolinium-containing agents as well as those with a severe atopic history or history of renal impairment. There are no known cases of NSF in patients with normal renal function(1). We will measure renal function in all patients within 1 month of the study.

For patients being scanned specifically for the study, we will select patients over 8 years of age, to avoid the need for general anaesthetic. We will attempt to select mainly patients who require MRI scanning with contrast for clinical indications. The control group will only consist of those having MRI for clinical indications. In this case, the only burden will be increased time in the scanner of around 20 minutes to obtain the sequences required. Evidence from our institution shows that the increased duration of general anaesthetic is not harmful and does not lead to complications or adverse events.

We will obtain blood samples for serum bio-marker measurement and haematocrit at the time of IV line insertion so this does not represent an additional intervention for the patient. We will use local anaesthetic cream or spray as requested by the patient and will use play and distraction techniques to minimise distress.

There are no potential adverse effects of a properly conducted transthoracic echocardiogram.

The 6 minute walk test will only be employed if the patient is able and willing to participate.

There are no potential adverse effects of a properly conducted MRI scan. The magnetic field and RF pulses are not known to cause any physical harm in properly selected subjects. Such selection will involve careful screening of the patients' medical history for any surgery or accidents that might have introduced metal to their bodies e.g. cerebral artery aneurysm clips or a metal foreign body in an eye. This will require a review of the patient's notes once consent has been given and a written checklist at the time of MRI scan. Such patients are not scanned in standard clinical practice and would also be excluded from the study.

Therefore, there is no realistic potential for pain, discomfort, distress, inconvenience or detrimental change to lifestyle anticipated for the participants from the MRI scan itself.

1. Dillman, J.R., J.H. Ellis, R.H. Cohan, P.J. Strouse, and S.C. Jan, Frequency and severity of acute allergic-like reactions to gadolinium-containing i.v. contrast media in children and adults. AJR Am J Roentgenol, 2007. 189(6): p. 1533-8.

Unexpected clinical findings

If new abnormalities or medical issues come to light as a result of the study investigations, the patient's GP and hospital consultant will be informed. Medical follow-up of these issues will be through the patient's usual medical carers.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of DCM for 3 months
* Ability to cooperate with MRI scan without general anaesthesia (volunteers over 8 years), or any age if cardiac MRi clinically indicated
* Provides written, informed consent

Exclusion Criteria:

* Patient exclusion criteria:
* Estimated GFR <30mls/min
* Contraindication to MRI (see appendix 1)
* Chronic inflammation/ malignancy/ connective tissue disease
* Structural congenital heart disease/ previous cardiac surgery

Control Group Exclusion Criteria:

* History of heart failure or congenital heart disease
* Contraindication to MRI (see below)
* Chronic inflammation/ malignancy/ connective tissue disease
* Previous malignancy

Exclusion criteria for MRI

* Central nervous system aneurysm clips
* Implanted neural stimulator
* Implanted cardiac pacemaker or defibrillator
* Cochlear implant
* Ocular foreign body e.g. metal shavings
* Other implanted medical devices e.g. drug infusion ports
* Insulin pump
* Metal shrapnel or bullet
* Pregnant women (patients who are uncertain will be required to have a urinary or blood screening test)

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Heart Failure Patients (MRI Clinically indicated)
  2. Heart Failure Patients (Voluntarily recruited from clinic)
     1. 8-16 years of age
     2. Non-GA only
  3. Control subjects (Clinically indicated brain MRI with contrast)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Estimated); Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Fibrosis | 6 months
  Higher fibrosis score (ECV) in heart failure patients in comparison to control subjects

SECONDARY OUTCOMES:
Biomarkers | 6 months
  Significantly different pattern of blood biomarkers in heart failure patients as compared to control subjects
Disease Severity | 6 months
  Significant correlation between fibrosis score on MRI or biomarker profile and clinical parameters (including 6 minute walk test and disease severity).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burch, MD, Study Director — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital NHS Trust, London, United Kingdom